CLINICAL TRIAL: NCT04244890
Title: Feasibility of Respiratory Management of Infants Needing Positive Pressure Ventilation or CPAP, Using a Single System to Deliver Uninterrupted Support Directly at Birth and the First Hours of Life
Brief Title: Feasibility of Uninterrupted Infant Respiratory Support Treatment
Acronym: FUIRST
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Drevhammar, Senior Consultant, PhD, Karolinska Institutet
Other Study IDs: 2019-05581
Record Dates: First submitted 2020-01-10; First posted 2020-01-28 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Respiratory Distress Syndrome, Newborn; Infant, Newborn; Respiratory Insufficiency Syndrome of Newborn
Keywords: Continuous Positive Airway Pressure; Resuscitation
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uninterrupted CPAP: Newborn infants in need of respiratory support directly after birth
  Interventions: Device: Uninterrupted CPAP for the first hours of life

INTERVENTIONS:
Device: Uninterrupted CPAP for the first hours of life — Directly at birth the infant will be supported with PPV with PEEP as needed, followed by nasal CPAP. Support will be provided with a single device for up to four hours.

SUMMARY:
Feasibility study of a simplified respiratory support system for newborn infants

DETAILED DESCRIPTION:
The study is a "proof-of-concept" feasibility trial that evaluates usage of a simplified respiratory support system for newborn infants. The study aims to evaluate both the feasibility of providing uninterrupted support for the first hours of life as well as a modified respiratory support system.

The system is a modified version of the commercially available rPAP system. The revised design has a simplified gas supply and allows elimination of a complicated driver. The new system has low resistance to breathing equal to the rPAP system. The study will recruit 40-60 infants in a single centre without a comparison arm.

The trial is conducted as a first step towards a large randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery at gestational age between 28+0 and 34+6
* Caesarean section at gestational age between 28+0 and 37+6
* Infants in need of respiratory support in delivery-room

Exclusion Criteria:

* Carciac malformations
* Airway malformations
* Known syndromes or neuromuscular disorders
* Transfer to other hospital within 4 hours likely

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborn infants in need of respiratory support directly after birth. Consent will be obtained from parents before delivery. Infants will be enrolled when investigators are available (convenience sample).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Number of interruptions in CPAP treatment | 0-240 minutes
  Number of CPAP-support interruptions (n)
Duration of interruptions in CPAP treatment | 0-240 minutes
  Duration CPAP support interruptions (min)
Cause of each interruption in CPAP treatment | 0-240 minutes
  Reported reason for interruptions in CPAP treatment (free text as reported by staff)

SECONDARY OUTCOMES:
Ease of use: Respiratory support system set up | 0-10 minutes
  How easy was the system to set up? (Easy/Minor problems/Major difficulties)
Ease of use: Airway and respiratory supportmanagement | 0-60 minutes
  How easy was airway and respiratory support management with the new system? (Easy/Minor problems/Major difficulties)
Ease of use: Fixation and transport | 0-60 minutes
  How easy was fixation and transport from the delivery room? (Easy/Minor problems/Major difficulties)
Level of respiratory support | 0-240 minutes
  What level of respiratory support was required? (Need for PPV, FiO2 and CPAP level)
Response to respiratory support | 0-240 minutes
  How did the infant respond to the given respiratory support? (SpO2, PaCO2, Temperature)
Respiratory support at 48 hours | 0-240 minutes
  What respiratory support did the infant receive at 48 hours of age
Rare events in clinical management | 0-240 minutes
  Did any infant need chest compression, intubation or any other rare interventions?
Adverse events and safety | 0-240 minutes
  Was there any suspected or confirmed adverse events related to equipment or the research protocol?

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Drevhammar, PhD, Study Director — meaning.....
Locations (1):
- Karolinska University Hospital, Neonatology department, Stockholm, Sweden

REFERENCES:
- [Derived] Baldursdottir S, Gunnarsdottir K, Donaldsson S, Jonsson B, Drevhammar T. Skin-to-skin stabilisation and uninterrupted respiratory support for preterm infants after birth: feasibility of a new and simplified rPAP system. Arch Dis Child Fetal Neonatal Ed. 2024 Oct 18;109(6):638-642. doi: 10.1136/archdischild-2023-326409. PMID 38514168